CLINICAL TRIAL: NCT00912002
Title: A Study to Investigate the Absorption, Metabolism, Excretion and Mass Balance After Administration of a Single Dose of [14C]MK-0941
Brief Title: A Study of Absorption, Metabolism, Excretion and Mass Balance After a Single Dose Administration of MK-0941 (MK-0941-016)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0941-016; 2008_598
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-0941 (Experimental): MK-0941
  Interventions: Drug: MK-0941

INTERVENTIONS:
Drug: MK-0941 — A single dose of 40 mg of [14C]MK-0941 (160 µCi), taken orally as eight 5-mg capsules

SUMMARY:
A single dose, open label study to characterize the routes of elimination and determine the mass balance of MK-0941. A single 40 mg dose of MK-0941 will be given orally to male participants with type 2 diabetes. After drug administration, blood, urine, and fecal samples will be collected to determine relative quantities of 14C-labeled MK-0941.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with type 2 diabetes, and is being treated with diet and exercise or with an oral anti-hyperglycemic agent
* Subject is willing to follow the American Heart Association diet and exercise program throughout the study
* Subject is a nonsmoker and/or has not used nicotine products for at least 6 months

Exclusion Criteria:

* Subject has a history of stroke, seizures, or major neurological disorder
* Subject has a history of neoplastic disease
* Subject has recently had abnormal bowel habits, such as diarrhea, loose stools or constipation
* Subject has a history of type 1 diabetes mellitus
* Subject has received insulin within the past 12 weeks
* Subject has a recent history of eye infection
* Subject has been diagnosed with glaucoma or is blind
* Subject consumes more than 3 alcoholic beverages per day
* Subject consumes more than 6 servings of coffee, tea, cola per day
* Subject has had major surgery, donated or lost blood in the past 4 weeks
* Subject has multiple or severe allergies to any food or drugs

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0941: Oral administration of a single 40-mg dose of [^14C]MK-0941 (160 µCi) to adult male subjects with type 2 diabetes.
Period: Overall Study
Arm/Group | MK-0941
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MK-0941
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  <29 years | 0
  29 years to 55 years | 6
  >55 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent of Dose Recovered in Urine and Feces Following a Single Oral Dose of [^14C]MK-0941 (160 µCi).
Description: Urine was collected at predose, 0 to 4, 4 to 8, 8 to 12, and 12 to 24 hr postdose, and at 24 hr intervals through subject discharge. Feces were collected at pre-dose and at 24 hr intervals through subject discharge. Subjects were discharged when the total recovery in urine and feces ≥90% of the administered dose or the recovery in urine and feces for two consecutive 24-hr intervals was ≤ 1%.
Time Frame: Up to 168 hours after study drug administration
Population: All treated participants.
Measure: Mean (Standard Deviation); unit: Percent Recovered
Groups:
- MK-0941: Oral administration of a single 40-mg dose of [^14C]MK-0941 (160 µCi) to adult male subjects with type 2 diabetes as eight 5-mg capsules.
Arm/Group | MK-0941
Number analyzed (Participants) | 6
Percent Recovered
  In the Urine | 60.0 (8.56)
  In the Feces | 38.7 (8.35)

2. Secondary Outcome: Number of Participants Who Experienced An Adverse Event
Time Frame: Up to 14 days after study drug administration
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | MK-0941
Number analyzed (Participants) | 6
participants | 5

3. Secondary Outcome: Number of Participants Who Discontinued the Study Due to An Adverse Event
Time Frame: Up to 14 days after study drug administration
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | MK-0941
Number analyzed (Participants) | 6
participants | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days after study drug administration
Arm/Group | MK-0941
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0941 (N=6)
Cataract (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Mucosal dryness (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.